CLINICAL TRIAL: NCT03923192
Title: Evaluation of Validity of the Near-infrared Imaging System (VistaCam iX Proxi) in Comparison With Digital Radiographic Findings and ICDAS-II in Detection of Approximal Carious Lesions: Diagnostic Accuracy Study.
Brief Title: Evaluation of Reliability of the Near-infrared Imaging System (VistaCam iX Proxi) in Comparison With Digital Radiographic Findings and ICDAS-II in Detection of Approximal Carious Lesions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Abdel Fattah Mahmoud Edrees, assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2411
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Proximal Dental Caries

STUDY DESIGN:
Intervention Model Description: screening of the Patients who join the Conservative Dentistry Department clinic will be done until the target population is achieved. The Patients' teeth will be subjected to visual examination and diagnosis using dental charts. once the patient is eligible to be included in this study, they will be contacted by the research investigator who will explain the study and identify the patient interests .If the patient show interest ,further clarification and discussing wil be held .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICDAS II (Other): Visual tactile examination based on ICDASII scoring system
  Interventions: Device: Vistacam; Radiation: Bitewing radiograph

INTERVENTIONS:
Device: Vistacam — device for early proximal caries detection
Radiation: Bitewing radiograph — radiograph for proximal caries detection

SUMMARY:
The aim of this study is to evaluate the Clinical performance of the near-infrared imaging system VistaCam iX Proxi in comparison with digital radiographic findings and ICDAS-II in detection of approximal carious lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 40 years.
* No gender restriction.
* Patients should have an acceptable oral hygiene level.
* Patients must have at least one posterior proximal caries

Exclusion Criteria:

* Patients with a compromised medical history.
* Severe or active periodontal disease.
* Heavy bruxism or a traumatic occlusion.
* Acute or chronic dental infection.
* Pregnant or breastfeeding women.
* Patients with posterior restorations on molars or premolars

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
dental caries | through study completion, an average of 1 year
  hidden proximal caries

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Other, Egypt

IPD SHARING:
Plan to Share IPD: Undecided